CLINICAL TRIAL: NCT03251651
Title: The Incidence of Postoperative Delirium According to the Different Intraoperative Sedatives, Dexmedetomidine vs. Propofol, in Elderly Patients Undergoing Orthopedic Lower Limb Surgery With Spinal Anesthesia: A Randomized Trial
Brief Title: Intraoperative Sedatives and Postoperative Deilirium
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Bundang Hospital (Other)
Responsible Party: Principal Investigator, Hyo-Seok Na, Associate Professor, Seoul National University Bundang Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: B-1704/391-304
Record Dates: First submitted 2017-08-14; First posted 2017-08-16 (Actual); Last update posted 2022-07-11 (Actual); Status verified 2022-07

CONDITIONS: Lower Extremity Problem; Delirium; Propofol; Dexmedetomidine
MeSH Terms: conditions — Delirium | interventions — Propofol; Dexmedetomidine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PPF (Experimental): Patient who received propofol during the operation
  Interventions: Drug: Propofol
- DEX (Experimental): Patient who received dexmedetomidine during the operation
  Interventions: Drug: Dexmedetomidine

INTERVENTIONS:
Drug: Propofol — Propofol is infused continuously via the target-controlled infusion device (Orchestra®, Fresenius vial, Brezins, France), and the effect-site concentration is maintained within 0.5-2.0 μg/ml.
  Arms: PPF
Drug: Dexmedetomidine — Dexmedetomidine is diluted with 0.9% saline to make a concentration of 4 μg/ml. As a loading dose, 1 μg/kg dexmedetomidine is administered over a 10-min period, which is then administered continuously at 0.1-0.5 μg/kg/h.
  Arms: DEX

SUMMARY:
Delirium occurs commonly in elderly patients. Its incidence after orthopedic surgery has been reported to be 5-61%. Delirium is classified into three sub-types: Hypoactive, hyperactive, and mixed. Although hyperactive delirium is not as common as hypoactive delirium, the abnormal behavior pattern of hyperactive delirium, such as agitation, confusion, or aggressiveness, is considered to be harmful to patients and medical personnel. Thus, it is important to promptly manage such behaviors associated with hyperactive delirium. Intraoperative sedation plays an important role in relieving anxiety or stress response of patients. Propofol-a common sedative agent-was reported to cause delirium more frequently, compared with dexmedetomidine, in post-cardiac surgery patients or mechanically-ventilated patients in the intensive care unit (ICU). In addition to the benefits of reducing opioid consumption and postoperative nausea/vomiting, dexmedetomidine is most often used for ICU sedation or procedural sedation. However, there has not been any prospective randomized study investigating how intraoperative dexmedetomidine sedation during regional anesthesia affects postoperative consciousness, perception, memory, behavior, emotion, and so on. In this study, based on the hypothesis that intraoperative dexmedetomidine sedation may reduce the incidence of abnormal psycho-motor behavior compared with propofol sedation, investigators prospectively will investigate the incidence of postoperative delirium in elderly patients who undergo orthopedic surgery with regional anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* Patients who undergo orthopedic surgery under spinal anesthesia
* Patients who want to sedation during the surgery
* Age of 65 years or greater
* American Society of Anesthesiologists physical status classification 1 and 2

Exclusion Criteria:

* General anesthesia
* Age < 65 years
* Patients who do not want to sedation during the surgery
* Patients who do not receive patient controlled analgesia postoperatively.
* Cognitive disorders
* Central nervous system disease, including dementia and Parkinson's disease

Ages: 65 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 748 (Actual)
Dates: Start 2017-06-15 (Actual); Primary Completion 2021-10-15 (Actual); Study Completion 2021-10-15 (Actual)

PRIMARY OUTCOMES:
Postoperative delirium | Within 3 day postoperatively
  The incidence of postoperative delirium

SECONDARY OUTCOMES:
Numerical rating scale | Postoperative 24 hour
  Postoperative pain score
Numerical rating scale | Postoperative 48 hour
  Postoperative pain score
Numerical rating scale | Postoperative 72 hour
  Postoperative pain score
Patient controlled analgesia (PCA) | Postoperative 24 hour
  Amounts of the PCA consumption
Patient controlled analgesia (PCA) | Postoperative 48 hour
  Amounts of the PCA consumption
Patient controlled analgesia (PCA) | Postoperative 72 hour
  Amounts of the PCA consumption
Rescue analgesics | Postoperative 24 hour
  Amounts of the analgesics administered to manage the postoperative pain
Rescue analgesics | postoperative 48 hour
  Amounts of the analgesics administered to manage the postoperative pain
Rescue analgesics | Postoperative 72 hour
  Amounts of the analgesics administered to manage the postoperative pain

CONTACTS AND LOCATIONS:
Overall Officials: Hyo-Seok Na, MD, PhD, Principal Investigator — Seoul National University Bundang Hospital
Locations (1):
- Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: No